CLINICAL TRIAL: NCT05777928
Title: Sleeve Gastrectomy and OverStitch™ Endoscopic Suturing System in the Modulation of Perceived Satiety
Brief Title: Bariatric Surgery and Modulation of Perceived Satiety
Acronym: BAR_SAZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43C102
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Obesity, Morbid
Keywords: obesity, satiety, Sleeve gastrectomy ,OverStitch
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve gastrectomy group (Experimental): Subjects with obesity candidates for sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy
- OverStitch™ Endoscopic Suturing System group (Experimental): Subjects candidates for a revision bariatric surgery with Overstitch endoscopic
  Interventions: Procedure: OverStitch™ Endoscopic Suturing System

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Sleeve gastrectomy involves vertical resection of a major part of the stomach, and a tubular remnant is retained along the lesser curvature.
  Arms: Sleeve gastrectomy group
Procedure: OverStitch™ Endoscopic Suturing System — Overstitch endoscopic procedure makes a review of gastro-jejunal anastomosis reducing surgical complications
  Arms: OverStitch™ Endoscopic Suturing System group

SUMMARY:
Bariatric surgery is the ideal therapeutic strategy for patients with severe obesity when lifestyle interventions have failed. Unfortunately, weight recovery after surgery affects one third of patients and is due to several factors, such as recovery of incorrect eating behaviour, reduction of physical activity or hormonal factors. Dilation of gastro-jejunal anastomosis is one of the main causes as it determines reduction of satiety in the patient and consequent increase of the portions of food consumed. In these cases it is necessary to make a review of gastro-jejunal anastomosis and to reduce surgical complications in recent years has been developed a method that allows the execution of sutures through a totally endoscopic way (OverStitch™ Endoscopic Suturing System).

Literature studies to assess hunger-satiety in patients undergoing bariatric surgery, suggest that surgery results in weight loss due to a series of changes in gastrointestinal physiology which impact on the feeling of hunger-satiety, and on the modification of the secretion of hormones involved in the regulation of gastric emptying such as the reduction of ghrelin secretion and the increase in postprandial cholecystokinin and GLP-1. There are no data in the literature on satiety in patients in previous bariatric surgery with weight recovery secondary to dilation of the gastro-jejunal anastomosis.

There are various methods to assess satiety, most of which are invasive and difficult to perform in routine clinical settings. A recently proposed method to evaluate the perception of satiety and validated on healthy adults, is the Water Load Tests (WLTs). The test consists in making the subject drink a quantity of water until he feels "pleasantly" full. The volume of water ingested is a valid indicator of the subjective feeling of satiety.

The aim of yhe study is to assess perceived satiety (measured by Water Load Test) after intervention of Sleeve Gastrectomy or a revision surgery with OverStitch™ Endoscopic Suturing System in obese individuals suitable for bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* subjects who are eligible for sleeve gastrectomy according to the SICOB criteria
* subjects, previously undergoing Sleeve Gastrectomy or gastric bypass, who, for weight regain, have been scheduled for revision surgery with the OverStitch™ Endoscopic Suturing System

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in satiety evaluated by water load test | At baseline and 6 months after the surgery
  Change in volume of water ingested during water load test

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bertoli, MD, Study Chair — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy